CLINICAL TRIAL: NCT04396639
Title: A SINGLE COUNTRY, MULTICENTER, OPEN-LABEL AND NON-RANDOMIZED CLINICAL TRIAL WITH MOROCTOCOG ALFA (AF-CC) PROPHYLAXIS AND TREATMENT OF BLEEDING EPISODES IN PREVIOUSLY TREATED PATIENTS WITH MODERATE AND SEVERE HEMOPHILIA A FOR A DURATION OF 8 WEEKS
Brief Title: Moroctocog Alfa (AF-CC) for Prophylaxis and Treatment of Bleeding Episodes in Previously Treated Hemophilia A Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1831097; 2020-004570-21 (EudraCT Number)
Record Dates: First submitted 2019-11-26; First posted 2020-05-20 (Actual); Results first posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Fifty eligible male subjects will be enrolled in the treatment arm to receive Moroctocog alfa (AF-CC) until 24 exposure days (EDs) or a period of up to 8 weeks on treatment had occurred (whichever occurs first).
  Interventions: Biological: Moroctocog-alfa (AF-CC)

INTERVENTIONS:
Biological: Moroctocog-alfa (AF-CC) — Moroctocog-alfa (AF-CC) is indicated for the control and prevention of hemorrhagic episodes and for routine and surgical prophylaxis in patients with hemophilia A (congenital factor VIII deficiency or classic hemophilia).
  Other Names: Xyntha

SUMMARY:
Moroctocog-alfa (AF-CC) is indicated for the control and prevention of hemorrhagic episodes and for routine and surgical prophylaxis in patients with hemophilia A (congenital factor VIII deficiency or classic hemophilia). The current single country, multi-centric, open label, non-randomized pragmatic clinical trial is a post-approval study to fulfill the Central Drugs Standard Control Organization (CDSCO) request for supplementary information relating to the use of moroctocog-alfa (AF-CC) in Indian subjects with hemophilia A.

The primary objective of study is to study the safety of moroctocog alfa (AF-CC) when administered for prophylaxis with respect to incidence of FVIII inhibitor development. The secondary objectives are to evaluate the incidence of adverse events (AEs) and serious adverse events (SAEs) in subjects receiving moroctocog alfa (AF-CC) prophylaxis, to evaluate the efficacy of moroctocog alfa (AF-CC) during a prophylaxis regimen, to evaluate the total annualized consumption of moroctocog alfa (AF-CC) by subjects following a prophylaxis regimen, to evaluate the efficacy of moroctocog alfa (AF-CC) for the treatment of breakthrough bleeding episodes (on-demand treatment) while following a prophylaxis regimen.

Fifty male subjects aged >/= 12 years to ≤65 years with moderate or severe hemophilia A will be enrolled in the study. The subjects will be selected based on protocol specified eligibility criteria. The overall treatment duration for each subject will be up to 8 weeks, with up to a 4-week screening period and a subsequent post-treatment 28-day safety observation period. Subjects are requested to continue in the study until 24 exposure days (EDs) or a period of up to 8 weeks on moroctocog alfa (AF-CC) treatment had occurred (whichever occurs first). Efficacy and safety assessments will be performed as specified in the protocol.

DETAILED DESCRIPTION:
Moroctocog-alfa (AF-CC) is indicated in India for the control and prevention of hemorrhagic episodes and for routine and surgical prophylaxis in patients with hemophilia A (congenital factor VIII deficiency or classic hemophilia). The current protocol outlines a post-approval study to fulfill the Central Drugs Standard Control Organization (CDSCO) written request for supplementary information relating to the use of moroctocog-alfa (AF-CC) in Indian subjects with hemophilia A. The additional information will include safety and efficacy of moroctocog-alfa (AF-CC) in Indian subjects with a diagnosis of congenital moderate or severe hemophilia A (FVIII:C ≤5%). The primary objective is to study the safety of moroctocog alfa (AF-CC) when administered for prophylaxis with respect to incidence of FVIII inhibitor development. The secondary objectives are to evaluate the incidence of adverse events (AEs) and serious adverse events (SAEs) in subjects receiving moroctocog alfa (AF-CC) prophylaxis, to evaluate the efficacy of moroctocog alfa (AF-CC) during a prophylaxis regimen, to evaluate the total annualized consumption of moroctocog alfa (AF-CC) by subjects following a prophylaxis regimen and to evaluate the efficacy of moroctocog alfa (AF-CC) for the treatment of breakthrough bleeding episodes (on-demand treatment) while following a prophylaxis regimen. The primary endpoint will be the proportion of subjects who develop FVIII inhibitor (≥0.6 BU/mL), as confirmed by central laboratory testing, during the course of the study. The secondary endpoints include assessment of incidence of AEs, incidence of SAEs, Annualized bleeding rate (ABR) during prophylaxis, Annualized total factor consumption (TFC) in international units (IU) and annualized TFC by weight (IU/kg) of moroctocog alfa (AF-CC) measured during the up to 8 weeks of treatment, by reason for infusion and total units consumed (across all reasons) and number of moroctocog alfa (AF-CC) infusions used to treat each bleed.

This study is a single-country, multicenter, open-label, interventional study which will be conducted in India. At least 50 male subjects aged ≥12 years to ≤65 years with moderate or severe hemophilia A (FVIII:C ≤5%) who have had at least 50 exposure days (EDs) to FVIII-containing products will be enrolled in the study. The overall treatment duration for each subject will be up to 8 weeks, with up to a 4-week screening period and a subsequent post-treatment 28-day safety observation period. Subjects are requested to continue in the study until 24 exposure days (EDs) or a period of up to 8 weeks on moroctocog alfa (AF-CC) treatment had occurred (whichever occurs first). Subjects will be treated with a dose and regimen of prophylaxis in accordance with the Local Product Development.

The following subjects will be included in this study:

1. Male subjects ≥12 years to ≤65 years with a diagnosis of congenital moderate or severe hemophilia A (FVIII:C ≤5%).
2. Documented history of at least 50 exposure days (EDs) to FVIII-containing products.
3. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative, parent(s)/legal guardian) has been informed of all pertinent aspects of the study. For minors under the age of legal consent in India, assent of the participating child needs to be documented for the age range 12 to 18 in addition to the parental informed consent.

Subjects presenting with any of the following will not be included in the study:

1. Prior history of inhibitor to FVIII or positive inhibitor testing (≥0.6 BU/mL) during Screening. Clinical signs or symptoms of decreased response to FVIII.
2. Known hypersensitivity to the active substance or any of the excipients.
3. Known allergic reaction to hamster proteins.
4. Presence of any bleeding disorder in addition to hemophilia A.
5. Participation in other studies involving investigational drug(s) (Phases 1-4) within 30 days before the current study begins and/or during study participation.
6. Planned surgery within 6 months from the start of the study.
7. Unsuitable to participate in study for any other reason as assessed by the investigator; including any disorder, except for conditions associated with hemophilia A, which in the investigator's opinion might jeopardize subject's safety or compliance with the protocol.
8. Subjects (or a legally acceptable representative) is not able to understand study documents and study procedure.
9. Immunocompromised subjects due to human immunodeficiency virus (HIV) infection (defined as viral load above or equal to 100,000 copies/mL; and for HIV+ subjects: cluster of differentiation 4 positive (CD4+) lymphocyte count below or equal to 200/μL). HIV status and CD4+ lymphocyte count results may be obtained at screening or from available medical records; results must be not older than 6 months prior to screening.
10. Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, subjects who have been previously enrolled into the study, or subjects who are Pfizer employees directly involved in the conduct of the study.
11. Planned use of any non-study medication for treatment of hemophilia (eg, other factor replacement agents, bypassing agents, or non-factor treatments [such as anti-tissue factor pathway inhibitors]).

The investigator will assign subject identification numbers sequentially to the subjects as they are screened for the study. This identification number will be retained throughout the study. Pfizer will provide the investigators with a sufficient amount of moroctocog alfa (AF-CC). Once moroctocog alfa (AF-CC) is dispensed to a subject it must not be re-dispensed to another subject. The product should be prepared, reconstituted, and used in accordance with procedures provided by their physicians. Moroctocog alfa (AF-CC) will be administered by the investigator or a delegate at Visits 2 and 3. For administration between study visits, the product will be administered in accordance with procedures provided by their physicians. Subjects or caregivers/parents of subjects will be trained on how to administer moroctocog alfa (AF-CC) away from the study site, as applicable. Moroctocog alfa (AF-CC) should be administered prophylactically in previously treated patients at a dose of 30±5 IU/kg given 3 times weekly. For on-demand treatment, the amount to be administered and the frequency of administration should always be tailored to the clinical effectiveness in individual subjects. In the interest of simplifying dosing and minimizing potential waste, a dosing variance of ±5 IU/kg is permitted throughout the study.

The investigator, or an approved representative, eg, study coordinator, will ensure that all investigational products, including any comparative agents and/or marketed products are stored in a secured area with controlled access under recommended storage conditions and in accordance with applicable regulatory requirements. Moroctocog alfa (AF-CC) should be stored in its original container and in accordance with the storage conditions stated on the label. The reconstituted solution of moroctocog alfa (AF-CC) may be stored at room temperature prior to infusion. The reconstituted solution of moroctocog alfa (AF-CC) does not contain preservative and should be infused within 3 hours after reconstitution. The investigator's site must maintain adequate records documenting the receipt, use, loss, or other disposition of the drug supplies. When investigational product is taken home by the subject, any unused products must be returned to the investigator by the subject at Visit 4. All used and unused vials of moroctocog alfa (AF-CC) and unused diluent syringes will be used for investigational product accountability. Administration of moroctocog alfa (AF-CC) by subjects or their caregivers away from the study site should be captured in the Subject Infusion Log. The monitor will review drug accountability during routine monitoring visits. Drug accountability will be done at all study visits after Day 1 until Visit 4. Any discrepancies must be investigated and their resolution documented.

The use of permitted concomitant medication must be in accordance with the study drug label. The use of concomitant treatments will be recorded throughout the study.

Study visits will include screening visit( Visit 1- within 28 Days prior to Day 1), Visit 2 (Day 1), Visit 3 (Day 24-32), Visit 4(Day 52-60) and End of Study Visit (Day 80-88 or earlier) Subjects may withdraw from the study at any time at their own request, or they may be withdrawn at any time at the discretion of the investigator. Any subject who uses non-study medication for the treatment of hemophilia (eg, other factor replacement agents, bypassing agents, or non-factor treatments [such as anti-tissue factor pathway inhibitors]) will be considered to have a protocol violation and will be withdrawn from the study. The exception to this would be for subjects who require non-study treatment for a bleed away from the study site. This would be considered a protocol deviation rather than a protocol violation that would not require withdrawal from the study. Subjects will be withdrawn from the study if their central laboratory result for inhibitor assessment at screening does not confirm eligibility per the local laboratory result.

The safety assessments throughout the study will include collection of AEs, laboratory safety testing, vital signs, and physical examination at the time points specified in protocol, but can be conducted at other time points at the investigator's discretion. All observed or volunteered AEs regardless of suspected causal relationship to the investigational product(s) will be reported as described in the protocol. The efficacy assessments include Total Factor VIII Consumption and bleeds including, Annualized Bleeding Rate During Prophylaxis, Number of Moroctocog alfa (AF-CC) Infusions Used to Treat Each Bleed, Annualized Total Factor Consumption of Moroctocog Alfa (AF-CC). All data will be collected in the case report form.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects ≥12 years to ≤65 years with a diagnosis of congenital moderate or severe hemophilia A (FVIII:C ≤5%).
2. Documented history of at least 50 exposure days (EDs) to FVIII-containing products.
3. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative, parent(s)/legal guardian) has been informed of all pertinent aspects of the study. For minors under the age of legal consent in India, assent of the participating child needs to be documented for the age range 12 to 18 in addition to the parental informed consent.

Exclusion Criteria:

1. Prior history of inhibitor to FVIII or positive inhibitor testing (≥0.6 BU/mL) during Screening. Clinical signs or symptoms of decreased response to FVIII.
2. Known hypersensitivity to the active substance or any of the excipients.
3. Known allergic reaction to hamster proteins.
4. Presence of any bleeding disorder in addition to hemophilia A.
5. Participation in other studies involving investigational drug(s) (Phases 1-4) within 30 days before the current study begins and/or during study participation.
6. Planned surgery within 6 months from the start of the study.
7. Unsuitable to participate in study for any other reason as assessed by the investigator; including any disorder, except for conditions associated with hemophilia A, which in the investigator's opinion might jeopardize subject's safety or compliance with the protocol.
8. Subjects (or a legally acceptable representative) is not able to understand study documents and study procedure.
9. Immunocompromised subjects due to human immunodeficiency virus (HIV) infection (defined as viral load above or equal to 100,000 copies/mL; and for HIV+ subjects: cluster of differentiation 4 positive (CD4+) lymphocyte count below or equal to 200/μL). HIV status and CD4+ lymphocyte count results may be obtained at screening or from available medical records; results must be not older than 6 months prior to screening.
10. Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, subjects who have been previously enrolled into the study, or subjects who are Pfizer employees directly involved in the conduct of the study.
11. Planned use of any non-study medication for treatment of hemophilia (eg, other factor replacement agents, bypassing agents, or non-factor treatments [such as anti-tissue factor pathway inhibitors]).

    -

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2020-01-25 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- India (5):
  - Nirmal Hospital, Surat, Gujarat
  - K.J.Somaiya Hospital and Research Centre, Mumbai, Maharashtra
  - Sahyadri Clinical Research and Development Centre, Pune, Maharashtra
  - Sahyadri Super Specialty Hospital, Pune, Maharashtra
  - Christian Medical College and Hospital, Ludhiana, Punjab

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1831097

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study, participants aged greater than or equal to (>=) 12 years to less than or equal to (<=) 65 years, with moderate or severe hemophilia A (circulating factor VIII [FVIII: C] <=5 percent [%]), who previously had at least 50 exposure days to FVIII-containing products were enrolled.
Groups:
- Moroctocog Alfa (AF-CC): Moroctocog alfa was administered prophylactically at a dose of 30 international unit per kilogram (IU/kg), 3 times weekly in accordance with local product document and with procedures provided by physicians. For on-demand treatment, the amount administered and the frequency of administration of moroctocog alfa was tailored to the clinical effectiveness in individual participants by their physicians. Participants continued participating in the study until 24 exposure days or until 8 weeks of treatment (whichever occurred first). Post treatment participants were followed up to 28 days.
Period: Overall Study
Arm/Group | Moroctocog Alfa (AF-CC)
Started | 50
Completed Follow up | 48
Completed | 48
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of moroctocog alfa.
Groups:
- Moroctocog Alfa (AF-CC): Moroctocog alfa was administered prophylactically at a dose of 30 IU/kg, 3 times weekly in accordance with local product document and with procedures provided by physicians. For on-demand treatment, the amount administered and the frequency of administration of moroctocog alfa was tailored to the clinical effectiveness in individual participants by their physicians. Participants continued participating in the study until 24 exposure days or until 8 weeks of treatment (whichever occurred first). Post treatment participants were followed up to 28 days.
Arm/Group | Moroctocog Alfa (AF-CC)
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.58 (9.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 50
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Developed Factor VIII (FVIII) Inhibitors
Description: FVIII inhibitor development was defined as an inhibitor titer of >=0.6 Bethesda units per milliliter (BU)/mL as confirmed by the central laboratory during the course of the study.
Time Frame: 24 exposure days or 8 weeks of treatment during the study (whichever occurred first)
Population: Safety analysis set included all participants who received at least 1 dose of moroctocog alfa.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Moroctocog Alfa (AF-CC)
Number analyzed (Participants) | 50
percentage of participants | 0 [0.00 to 0.06]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. In this outcome measure all AEs are reported.
Time Frame: Day 1 up to 28 days after last dose of study drug (approximately maximum up to 12 Weeks)
Population: Safety analysis set included all participants who received at least 1 dose of moroctocog alfa.
Measure: Count of Participants; unit: Participants
Arm/Group | Moroctocog Alfa (AF-CC)
Number analyzed (Participants) | 50
Participants | 3

3. Secondary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (SAEs)
Description: SAEs: an adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; inpatient hospitalization or prolongation of existing hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect. Treatment emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Day 1 up to 28 days after last dose of study drug (approximately maximum up to 12 Weeks)
Population: Safety analysis set included all participants who received at least 1 dose of moroctocog alfa.
Measure: Count of Participants; unit: Participants
Arm/Group | Moroctocog Alfa (AF-CC)
Number analyzed (Participants) | 50
Participants | 0

4. Secondary Outcome: Mean Annualized Bleeding Rate (ABR) During Prophylaxis
Description: Participants who had bleeding episode, ABR was derived by the following formula: ABR = number of bleeds per treatment interval duration per 365.25. Participants who did not have bleeding episodes, ABR was 0. In this outcome measure, mean ABR was reported considering all the participants (with bleeding episodes and without bleeding episodes).
Time Frame: 24 exposure days or 8 weeks of treatment during the study (whichever occurred first)
Population: Safety analysis set included all participants who received at least 1 dose of moroctocog alfa.
Measure: Mean (Standard Deviation); unit: bleed rate per year
Arm/Group | Moroctocog Alfa (AF-CC)
Number analyzed (Participants) | 50
bleed rate per year | 0.79 (2.042)

5. Secondary Outcome: Mean Annualized Total Factor Consumption (TFC)
Description: The total amount in international units (IU) infused for each infusion recorded were summed to calculate the TFC for each participant during the treatment interval duration (up to 8 weeks of treatment, or sooner, once 24 exposure days are achieved). The annualized TFC of moroctocog alfa was derived for each participant by using the following formula: Annualized TFC = (TFC / treatment interval duration)*365.25.
Time Frame: 24 exposure days or 8 weeks of treatment during the study (whichever occurred first)
Population: Safety analysis set included all participants who received at least 1 dose of moroctocog alfa.
Measure: Mean (Standard Deviation); unit: international units
Arm/Group | Moroctocog Alfa (AF-CC)
Number analyzed (Participants) | 50
international units | 287432.26 (93866.233)

6. Secondary Outcome: Mean Annualized Total Factor Consumption (TFC) by Weight
Description: The total amount in IU infused for each infusion recorded was summed to calculate the TFC for each participants during the treatment interval duration (up to 8 weeks of treatment, or sooner, once 24 exposure days are achieved). The annualized TFC of moroctocog alfa was derived for each participant by using the following formula: Annualized TFC = (TFC / treatment interval duration)*365.25. To calculate the annualized TFC per weight, the most recently recorded weight measurement was used.
Time Frame: 24 exposure days or 8 weeks of treatment during the study (whichever occurred first)
Population: Safety analysis set included all participants who received at least 1 dose of moroctocog alfa.
Measure: Mean (Standard Deviation); unit: international units per kilogram
Arm/Group | Moroctocog Alfa (AF-CC)
Number analyzed (Participants) | 50
international units per kilogram | 4175.67 (858.383)

7. Secondary Outcome: Mean Number of Moroctocog Alfa (AF-CC) Infusions Used to Treat Each New Bleed
Description: Number of moroctocog alfa infusions used to treat each bleed was calculated by adding the initial (on-demand) infusion to any subsequent (on-demand) infusions for the same bleed (same bleed start date/time). If there was more than one bleed location (e.g., ankle and joint) with identical bleed start date and time, it was treated as one bleed occurrence.
Time Frame: 24 exposure days or 8 weeks of treatment during the study (whichever occurred first)
Population: Safety analysis set included all participants who received at least 1 dose of moroctocog alfa. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: infusions per bleed
Units Other Than Participants: bleeds
Arm/Group | Moroctocog Alfa (AF-CC)
Number analyzed (Participants) | 7
Number analyzed (bleeds) | 7
infusions per bleed | 1.0 (0.00)

ADVERSE EVENTS:
Time Frame: Day 1 up to 28 days after last dose of study drug (approximately maximum up to 12 Weeks)
Description: Same event may appear as AE and SAEs, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis set included all participants who received at least 1 dose of moroctocog alfa.
Arm/Group | Moroctocog Alfa (AF-CC)
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 3/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moroctocog Alfa (AF-CC) (N=50)
Vertigo (Ear and labyrinth disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT04396639/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT04396639/SAP_001.pdf